CLINICAL TRIAL: NCT03180489
Title: Does Dapagliflozin Provide Additional Health Benefits To Dietary Counseling For Weight Loss?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christopher Bell (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Christopher Bell, Associate Professor, Colorado State University
Organization: Colorado State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 17-7147H
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin with dietary counseling (Experimental): Daily oral administration of dapagliflozin tablet with dietary counseling to promote weight loss.
  Interventions: Drug: Dapagliflozin Tablet
- Placebo with dietary counseling (Placebo Comparator): Daily oral administration of placebo tablet with dietary counseling to promote weight loss.
  Interventions: Drug: Placebo Tablet

INTERVENTIONS:
Drug: Dapagliflozin Tablet — Daily oral administration of dapagliflozin with dietary counseling to promote weight loss. Dapagliflozin 5 mg tablet will begin as one tablet per day for the first 14-days. In the absence of complications, side effects, or unfavorable reactions, the dose will then increase to two tablets for the remainder of the study.
  Other Names: Farxiga
  Arms: Dapagliflozin with dietary counseling
Drug: Placebo Tablet — Daily administration of placebo tablet with dietary counseling to promote weight loss. Matching placebo for dapagliflozin 5 mg tablet will begin as one tablet per day for the first 14-days. In the absence of complications, side effects, or unfavorable reactions, the dose will then increase to two tablets for the remainder of the study.
  Arms: Placebo with dietary counseling

SUMMARY:
Dapagliflozin is a medicine to treat diabetes. Its mechanism of action is via sodium-glucose co-transporter 2 (SGLT2) inhibition. In adults with diabetes, use of sodium-glucose co-transporter 2 inhibitors is associated with moderate weight (fat) loss, in addition to other health benefits, including decreased blood pressure, decreased inflammation, and decreased oxidative stress. It is unclear as to whether these health benefits are due to SGLT2 inhibition per se, or as a secondary effect of weight loss. We wish to compare the health benefits of dietary counseling for weight loss with and without concomitant use of an SGLT2 inhibitor.

DETAILED DESCRIPTION:
This is a randomized, prospective, placebo-controlled, double blind, repeated measures study. 50 overweight/obese adults (body mas index > 27.5 kg/m2) will be recruited for participation and randomly assigned to one of two 12 week treatments: (1) daily oral administration of Dapagliflozin with dietary counseling to promote weight loss; or, (2) daily oral administration of a placebo with dietary counseling to promote weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Aged 18-65 years.
* No known Type 2 Diabetes
* Body mass index greater than or equal to 27.5 kg/m^2
* Limited exercise participation (maximum of 3/week regularly scheduled activity sessions of < 30 minutes during the previous month).
* Completion of a screening visit consisting of medical history, physical examination, and 12-lead electrocardiogram and blood pressure assessment at rest and during incremental exercise to volitional exhaustion (Note: Subjects with abnormal screening values may be eligible if the results are not clinically significant, as judged by the investigator or medical monitor)
* Agree to abide by the study schedule and dietary restrictions and to return for the required assessments
* Women of childbearing potential must have negative pregnancy test and be using acceptable contraception

Exclusion Criteria:

* Evidence of clinically significant cardiovascular, respiratory, renal, hepatic, pulmonary, gastrointestinal, haematological, neurological, psychiatric, or other disease that may interfere with the objectives of the study or the safety of the subject, as judged by the investigator in agreement with the sponsor or medical monitor, have been hospitalized in the past 2 years as a result of these conditions, or are receiving pharmacological treatment for these conditions.
* Use of prescription drugs (see exceptions listed below) or herbal preparations in the 2 weeks before study commencement. Prior use of medication or herbal preparations in the 4 weeks before study commencement that are intended for weight-loss and/or sold/marketed as weight-loss products or may alter metabolism. Permitted Prescription Drugs: Birth Control, Less than a 7 day short course of antibiotics. Note: Rifampicin is not permitted. Other medicines, such as those for gastroesophageal reflux disease, depression, and Over The Counter analgesics and allergy medications,may be allowed, but will be approved on a case-by-case basis.
* Is currently enrolled in another clinical study for another investigational drug or has taken any other investigational drug within 30 days before the screening visit.
* Habitual and/or recent use (within 2 years) of tobacco.
* Being considered unsuitable for participation in this trial for any reason, as judged by the investigator or medical monitor.
* History of serious hypersensitivity reaction to Dapagliflozin.
* Severe renal impairment, end-stage renal disease, or dialysis.
* Pregnant or breastfeeding individual.
* Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal and/or alanine aminotransferase (ALT) >3x upper limit of normal.
* Total bilirubin >2.0 mg/dL (34.2 umol/L).
* Positive serologic evidence of current infectious liver disease including Hepatitis B viral antibody immunoglobulin M, Hepatitis B surface antigen and Hepatitis C virus antibody.
* Estimated Glomerular Filtration Rate <60 mL/min/1.73 m^2 (calculated by Cockcroft-Gault formula).
* History of bladder cancer.
* Recent cardiovascular events in a patient, including any of the following: acute coronary syndrome within 2 months prior to enrolment; hospitalization for unstable angina or acute myocardial infarction within 2 months prior to enrolment; acute stroke or trans-ischemic attack within two months prior to enrolment; less than two months post coronary artery revascularization; congestive heart failure defined as New York Heart Association class IV, unstable or acute congestive heart failure. Note: eligible patients with congestive heart failure, especially those who are on diuretic therapy, should have careful monitoring of their volume status throughout the study.
* Blood pressure at enrolment: Systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg.
* Blood pressure at randomization: Systolic blood pressure ≥165 mmHg and/or diastolic blood pressure ≥100 mmHg
* Individuals who, in the judgment of the medical monitor, may be at risk for dehydration.
* Individuals with a history of fragility fracture, or bone mineral density values reflective of risk for fracture (DEXA Z-score <or= to -2 in pre-menopausal women, and men <50, and T-score <or= to -1) will not be permitted to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bell, Ph.D., Principal Investigator — Colorado State University; Christopher Melby, Dr.P.H., Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Dept. of Health and Exercise Science, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
Started | 33 | 29
Completed | 25 | 25
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 5 | 7 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: meters] | 1.69 (0.08) | 1.67 (0.09) | 1.68 (0.08)
Body Mass [Mean (Standard Deviation); unit: kg] | 96.5 (15.6) | 93.8 (20.4) | 95.13 (18.0)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 33.5 (3.9) | 33.2 (5.6) | 33.4 (4.7)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 116 (8) | 112 (10) | 114 (9)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 69 (5) | 69 (8) | 69 (7)
Peak Oxygen Uptake [Mean (Standard Deviation); unit: ml/kg/min] | 22.2 (5.0) | 24.8 (5.6) | 23.5 (5.4)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dL] | 74.7 (6.9) | 76.1 (7.7) | 75.4 (7.3)
Fasting Insulin [Mean (Standard Deviation); unit: mU/L] | 6.9 (0.8) | 11.1 (3.5) | 9.0 (12.7)
Dietary Intake [Mean (Standard Deviation); unit: kcal/day] | 1819 (491) | 2187 (541) | 2003 (538)
Carbohydrate [Mean (Standard Deviation); unit: g/day] | 197 (59) | 246 (73) | 222 (69)
Fat [Mean (Standard Deviation); unit: g/day] | 77 (26) | 91 (28) | 84 (28)
Protein [Mean (Standard Deviation); unit: g/day] | 80 (25) | 85 (24) | 83 (24)
eGFR [Mean (Standard Deviation); unit: mL/min/173m2] | 154 (52) | 152 (54) | 153 (52)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Insulin Sensitivity at Week 12 Via Oral Glucose Tolerance Test
Description: Insulin sensitivity was estimated by measuring circulating insulin concentrations after a 12 hour fast and after ingesting 75 g of glucose. Insulin was measured 0, 30, 60, 90 and 120 minutes after glucose ingestion. Time point 0 minutes is reported below.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
Number analyzed (Participants) | 25 | 25
mU/L
  Baseline | 6.9 (0.8) | 11.1 (3.5)
  12 Weeks | 5.5 (0.7) | 6.5 (1.0)

2. Primary Outcome: Change From Baseline in Blood Pressure at Week 12
Description: Blood pressure was measured with an automatic machine at baseline. Numbers are reported as systolic/diastolic
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
Number analyzed (Participants) | 25 | 25
mmHg
  Systolic | 116 (10) | 112 (8)
  Diastolic | 69 (8) | 69 (5)

3. Primary Outcome: Change From Baseline in Perception of Satiety at Week 12
Description: Participants answered a satiety questionnaire before liquid meal primer, immediately post liquid meal primer, 60 minutes post liquid primer, immediately post breakfast buffet, 60 minutes, 120 minutes and 180 minutes post breakfast buffet. Responses how full do you feel right now? for 60 minutes post liquid meal primer ingestion are reported below. This was determined by using a visual analog scale. The left side of the analog scale represents a null answer (e.g. How full do you feel right now)? Answer 0: Not full at all. The right side of the line represented the strongest answer in the opposite direction (e.g. How full to you feel right now)? Answer 100: Extremely full. The length of the line is 100 mm, thus the scale ranges for all answers were 0-100. All values are reported as values between 0 and 100. If the answers to the fullness questions increased, this represented a decreased desire to eat.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 27 (16) | 21 (12)
  12 Weeks | 31 (18) | 28 (16)

4. Primary Outcome: Change From Baseline in Perception of Hunger at Week 12
Description: Participants answered a hunger questionnaire before liquid meal primer, immediately post liquid meal primer, 60 minutes post liquid primer, immediately post breakfast buffet, 60 minutes, 120 minutes and 180 minutes post breakfast buffet. Responses to how hungry do you feel right now? for 60 minutes post liquid meal primer ingestion are reported below. This was determined by using a visual analog scale. The left side of the analog scale represents a null answer (e.g. How hungry do you feel right now? Answer 0: Not hungry at all. The right side of the line represented the strongest answer in the opposite direction (e.g. How full to you feel right now)? Answer 100: Extremely hungry. The length of the line is 100 mm, thus the scale ranges for all answers were 0-100. All values are reported as values between 0 and 100. If the answers to the fullness questions increased, this represented an increased desire to eat.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 42 (25) | 53 (18)
  12 Weeks | 39 (20) | 53 (21)

5. Primary Outcome: Change From Baseline in Marker of Inflammation (High Sensitive C-reactive Protein) at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Data not collected
Population: Data not collected
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Change From Baseline in Marker of Inflammation (Tumor Necrosis Factor Alpha) at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Data not collected
Population: Data not collected
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Change From Baseline in Marker of Inflammation (Interleukin 6) at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: data not collected
Population: Data not collected
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Change From Baseline in Hunger Hormone Ghrelin at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: data not collected
Population: Data not collected
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Change From Baseline in Hunger Hormone Peptide Tyrosine Tyrosine at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: data not collected
Population: Data not collected
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Change From Baseline in Maker of Oxidative Stress (Oxidized Low Density Lipoprotein) at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Data not collected
Population: Data not collected
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Change From Baseline in Maker of Oxidative Stress (Low Density Thiobarbituric Acid Reactive Substances) at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Data not collected
Population: Data not collected
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Change From Baseline in Satiety Hormone Leptin at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Data not collected
Population: Data not collected
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Change From Baseline in Satiety Hormone Insulin at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Data not collected
Population: Data not collected
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the 12 week intervention period.
Description: Subjects were withdrawn are included in the Adverse Event data but are not included in the analysis of the Baseline Characteristics and the Outcome Measures data.
Arm/Group | Dapagliflozin With Dietary Counseling | Placebo With Dietary Counseling
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/29
Other Adverse Events (participants affected / at risk) | 28/33 | 23/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin With Dietary Counseling (N=33) | Placebo With Dietary Counseling (N=29)
Allergies (Immune system disorders) | 2 (2) | 3 (3)
Cold Symptoms (Infections and infestations) | 15 (22) | 13 (22)
Stomach Pain and Diarrhea (Gastrointestinal disorders) | 6 (10) | 5 (6)
Headache and Dizziness (General disorders) | 10 (19) | 9 (15)
Muscle Joint Soreness and Pain (Musculoskeletal and connective tissue disorders) | 9 (13) | 6 (7)
Urinary Disorders, Yeast Infections and PMS (General disorders) | 6 (7) | 7 (15)
Tooth Pain (General disorders) | 1 (1) | 0 (0)
Cold Sores (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vitamin D Deficiency (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1)
Anxiety Attack (General disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT03180489/Prot_SAP_ICF_000.pdf